CLINICAL TRIAL: NCT03589118
Title: Qi Gong as a Method of Craving Reduction in Severe Addict Patients
Acronym: QICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P160946J; 2017-A02986-47 (Registry Identifier: IDRCB)
Record Dates: First submitted 2018-05-18; First posted 2018-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Addiction; Alcohol Dependence
Keywords: Substance Addiction; Craving; Chinese Medecine; Qi Gong; Psychology
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Patients are randomized in two groups :
  * usual medical and psychological support in the control group
  * qi gong sessions added in the experimental group
  Allocation between groups qi and control is 1 : 1
Who Masked: Outcomes Assessor
Masking Description: Primary outcome (VAS scale) will be presented to the patient and reported by a study nurse blinded of the randomization arm of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qi Gong (Experimental): Qi gong sessions added to usual well defined medical and psychological support
  Interventions: Other: Qi Gong sessions
- Control (No Intervention): Usual well defined medical and psychological support

INTERVENTIONS:
Other: Qi Gong sessions — 13 sessions of Qi Gong in a 9 weeks period
  Arms: Qi Gong

SUMMARY:
Craving arises in response to an affective tone that is associated with perceptual representations of a sensory object, rather than directly in response to the object.

The investigators presume that qi gong functions to decouple pleasant and unpleasant experience from habitual reactions by removing the affective bias that fuels such emotional reactivity. Qi gong training may specifically target the associated learning process with an emphasis on the critical link between affect and craving in an addictive loop.

DETAILED DESCRIPTION:
The treatment of severe addiction to alcohol and one other or more psychoactive substances sometimes requires hospitalization for complex withdrawal. The medical term " sevrage complexe " is used in this file for hospitalization of patients with multiple addictions or with multiple comorbidities. In the french regulation the duration of hospitalization for " sevrage complexe " is at least 13 days.

The acute period of the first week is sufficient for physical weaning. A period relay for maintaining abstinence beyond the acute phase is a difficult stage. During this period the psychological craving related to the absence of the product causes dysphoria, stress, emotivity and increased difficulty in managing psychological aggression. The risk of relapse is then maximal and favored by many insults of everyday life.

Qi gong is classified by US National Library of Medicine as a mind-body therapy (MBT). It's an ancient traditional Chinese health practice believed to have special healing and recovery power. Today millions of people practice qi gong in China and around the world to treat various diseases. Qi gong is an ecole of breath, relaxation, guided imagery and inward attention. Practice of qi gong is believed to help cleanse the body of toxins, restore energy balance, reduce stress and anxiety. The Baduanjin qigong is one of the most common form of Chinese qi gong.

When going through withdrawal, craving is a psychological urge to administer a discontinued medication or recreational drug. Craving episodes may be triggered by seeing objects or experiencing moments that are associated with the drug or usage of it, and this phenomenon is termed post-acute withdrawal syndrome.

The main goal of our study is to demonstrate a reduction of craving during alcohol and coaddictions withdrawal. This demonstration is of first importance: first for the well-being of the patient during the first weeks after withdrawal, second for drug savings, and third abstinence rate because many authors consider that craving intensity is correlated with relapses risk.

The mind-body techniques of traditional Chinese medicine, as Qigong, are inscribed the number of current approaches in residential treatment. Their transmission would be an additional contribution to the stabilization via active management and motivated patient himself on his health.

The compulsion associated with addictive behavior can be defined as a pathological change in brain plasticity. The pathological learning process induced by the repeated use of the substance is causing behavioral control loss in the vulnerable individual.

Considering the impulsive nature of craving, this study will investigate the driving dynamics of impulses: Trieb "push". Return to the perception supported by the development of attention gestures leaning on the breath, puts us ahead of the motor action and is potentially a mean of influencing compulsive process.

ELIGIBILITY:
Inclusion criteria

* Meets DSM 5 criteria for alcohol use disorder and other substance use disorders
* Alcohol is one of the major abused substances if using multiple substances
* Severity of the disorder defines by the necessity of a complex withdrawal hospitalization.
* Used alcohol in the 3 weeks before hospitalization
* Seeks addiction treatment
* Patient willing to adhere to the study protocol (e.g. attend all visits and follow-ups in the next 3 months).
* Age ≥ 18
* Negative pregnancy test (βHCG) for women of child bearing potential
* Signed informed consent
* Affiliation to the French health insurance (recipient or assign)
* Oral and written comprehension of the french langage

Non-inclusion criteria

* Pose a current suicidal risk including active suicidal ideation and suicide attempt in the past 30 days
* Non stabilized severe psychiatric comorbidities such as bipolar disorder, schizophrenia, … (at the investigator's discretion)
* Pregnant or breastfeeding women
* Decompensated cirrhosis, liver encephalopathy, neurological complications, severe cognitive impairment and any other severe somatic comorbidity (at the investigator's discretion)
* Currently participated in other interventional clinical study
* Individuals placed under guardianship
* Patient deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Variation of craving intensity | Change in VAS from baseline to 9 weeks treatment
  Variation of craving intensity on a Vvisual aAnalogic sScale (VAS) between baseline and the end of the treatment. The intensity is measured by "not at all" (score of 0) and "craving as bad as it could be" or "the most I've ever felt " (maximum score of 10), self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents his craving intensity.
  The score is determined by measuring the distance on the 10-cm line between the "no craving" anchor and the patient's mark.

SECONDARY OUTCOMES:
Evolution over time of craving intensity | 0 day, 3 days, 5 days, 3 weeks and 9 weeks post-baseline
  Craving intensity measured with 14-items Obsessive Compulsive Drinking Scale (OCDS).
  OCDS score is the sum of two subscales scores. Obsessive Subscale is calculated from items 1 to 6, maximal subscore is 20 (worse outcome).
  Compulsive subscale is calculated from items 7 to 14.
Difference in treatment retention | 3 weeks and 9 weeks post-baseline
  Difference in treatment retention (permanence rate)
Evolution over time of total alcohol consumption | 0 day, 3 days, 5 days, 3 weeks and 9 weeks post-baseline
  Alcohol consumption assessed with Time Line Follow Back (TLFB)
Evoluation over time of anxiety | 0 day, 3 days, 5 days, 3 weeks and 9 weeks post-baseline
  Anxiety questions sum score of Hospital Anxiety and Depression scale (HAD scale). Seven questions are related to anxiety (total A). Anxiety is measured by the sum score questions 1 , 4, 6 , 8, 10 , 12, 14. . Non : Total A = 1,3,5,7,9,11,13
  The maximum score being equal to 21 :
  0-7: normal; 8-10 bordeline abnormal (borderline case); 11-21 : abnormal (case)
Evolution over time of depression | 0 day, 3 days, 5 days, 3 weeks and 9 weeks post-baseline
  Depression questions sum score of Hospital Anxiety and Depression scale (HAD scale).
  Seven questions are related to the depressive dimension (total D). Depression is measured by the sum score questions 2, 3, 5 , 7, 9 , 11, 13 Non: Total D : 2,4,6,8,10,12,14.
  The maximum score being equal to 21 :
  0-7: normal; 8-10: bordeline abnormal (borderline case); 11-21: abnormal (case)
Psycological qualitative evaluation | 1 day, 2 days, 3 days, 4 days, 5 days, 2 weeks, 3 weeks, 4 weeks, 5 weeks, 6 weeks, 7 weeks, 8 weeks and 9 weeks post-baseline
  Qualitative evaluation assessed with clinical notes
Evolution over time of total alcohol consumption measured by GGT biomarker | at 0 day, 3 days, 5 days, 3 weeks and 9 weeks post-baseline
  GGT Gamma glutamyl transpeptidase levels in UI/I
Evolution over time of total alcohol consumption measured by Carbohydrate-Deficient Transferrin (CDT) marker | at 0 day, 3 days, 5 days, 3 weeks and 9 weeks post-baseline
  CDT levels in %
Evolution over time of total alcohol consumption measured by Mean Globular Volume (MGV) marker | at 0 day, 3 days, 5 days, 3 weeks and 9 weeks post-baseline
  MGV levels in fL

CONTACTS AND LOCATIONS:
Overall Officials: Alain BAUMELOU, MD, Ph.D, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Nathalie PLET, Ph.D, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Saint ELOI, Montpellier
  - Hôpital L'ARCHET, Nice
  - Groupe Hospitalier Pitié Salpêtrière, Paris